CLINICAL TRIAL: NCT03671707
Title: A Combined Cessation Intervention of Brief Advice, Nicotine Replacement Therapy Sampling and Active Referral (BANSAR) for Smoking Fathers: a Multicenter, Single-blinded, Pragmatic Randomised Controlled Trial
Brief Title: Brief Advice, Nicotine Replacement Therapy Sampling and Active Referral (BANSAR) for Smoking Fathers
Acronym: BANSAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government); Queen Mary Hospital, Hong Kong (Other); Pamela Youde Nethersole Eastern Hospital (Other); Kwong Wah Hospital (Other); Queen Elizabeth Hospital, Hong Kong (Other); United Christian Hospital (Other); Princess Margaret Hospital, Hong Kong (Other Government); Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15162691; HKUCTR-2422 (Registry Identifier: HKU Clinical Trials Registry)
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Smoking Cessation; Tobacco Use Cessation
Keywords: tobacco dependence treatment; combined brief intervention; AWARD advice; active referral; nicotine replacement therapy; pregnancy; family health; Chinese
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation | interventions — corticosteroid hormone-induced factor; Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Brief AWARD advice + Nicotine replacement therapy sampling + Active referral
  Interventions: Behavioral: Brief AWARD advice; Drug: Nicotine replacement therapy sampling; Behavioral: Active referral
- Control group (Active Comparator): Very brief advice (VBA) + Leaflet
  Interventions: Behavioral: Very brief advice; Behavioral: Leaflet

INTERVENTIONS:
Behavioral: Brief AWARD advice — Subject will receive brief, face-to-face counselling following a structured AWARD model at baseline :
  1. Ask: smokers will be asked about their smoking behaviour
  2. Warn about the harms of smoking using a leaflet which contain information about harms of secondhand smoke to women, fetus and infant, motivational messages to quit and smoking cessation services.
  3. Advise to quit or reduce their smoking and use the provided 1-week nicotine replace therapy sample as soon as possible
  4. Refer smokers to smoking cessation services if they agree.
  5. Do-it-again: repeat the AWARD advise through telephone boosters at 2-week and 4-week after baseline
  Other Names: Ask, Warn, Advise, Refer and Do-it-again
  Arms: Intervention group
Drug: Nicotine replacement therapy sampling — Subjects will receive 1-week supply of free nicotine patch or gum with dosage based on participants' number of cigarette per day. An information card containing reminders of nicotine replacement therapy use and actions to handle potential side effects will be provided.
  Other Names: NRT sample
  Arms: Intervention group
Behavioral: Active referral — Subjects will be encouraged to select and access a smoking cessation services in Hong Kong. If the subjects agree, their contact information will be sent to the smoking cessation service providers for further arrangement.
  Arms: Intervention group
Behavioral: Very brief advice — Subjects will receive general advice to quit
  Other Names: VBA
  Arms: Control group
Behavioral: Leaflet — Subjects will receive a standard leaflet on perinatal smoking by Department of Health
  Other Names: Print-based material
  Arms: Control group

SUMMARY:
This study aims to evaluate the effects of a combined "cocktail", cessation intervention of brief advice, nicotine replacement therapy sampling and active referral (BANSAR) for smoking expectant fathers on smoking cessation outcomes

DETAILED DESCRIPTION:
Secondhand smoke (SHS) exposure cause substantial harms to pregnant women, foeti and infants. Smoking cessation (SC) interventions for smoking expectant fathers are needed particularly in China where male smoking predominates and many pregnant women (about 30% in Hong Kong) were exposed to SHS. Prenatal period presents a valuable teachable moment to engage smoking expectant father in tobacco dependence treatment. However, most smoking cessation trials were conducted in the Western countries on smoking pregnant women or smoking couples. Very few trials were designed to target fathers quitting.

Given the busy clinical settings in Hong Kong Public Hospitals, evidence-based, low-cost and sustainable brief cessation intervention applicable in real-world practice is imperative. Informed by previous research, a combined cessation intervention of brief advice, nicotine replacement therapy sampling and active referral (BANSAR) has been developed for smoking expectant father. This multicentre, pragmatic, assessor-blinded, individually-randomized controlled trial aims to evaluate BANSAR for smoking cessation outcomes in smoking expectant father visiting prenatal clinics in Hong Kong

ELIGIBILITY:
Inclusion criteria for both expectant father and mother:

1. Hong Kong resident aged 18 or above
2. Able to read and communicate in Chinese
3. Living together in the past 7 days

Inclusion criteria for expectant father:

1. Having smoked 1 or more cigarettes daily in the past 3 months
2. Having a telephone or mobile phone contact

Inclusion criteria for expectant mother:

1. Not having smoked any cigarette in the past 30 days

Exclusion Criteria for expectant father

1. Having any history of severe angina, arrhythmia, or acute myocardial infarction
2. Having psychiatric/psychological diseases or regular psychotropic medications
3. Having used smoking cessation aids or participated in other smoking cessation services or projects in the past 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Biochemically-validated abstinence | 6-month after baseline
  Defined by an exhaled carbon monoxide level of < 4 parts per million (ppm)

SECONDARY OUTCOMES:
Self-reported past 7-day abstinence | 3-month after baseline
  Being completely smoke-free in the past 7 days
Self-reported past 7-day abstinence | 6-month after baseline
  Being completely smoke-free in the past 7 days
Self-reported continuous abstinence in the past 24-week | 6-month after baseline
  Being completely smoke-free in the past 24-week
Smoking reduction | 3-month after baseline
  Defined by at least 50% reduction in baseline daily number of cigarettes
Smoking reduction | 6-month after baseline
  Defined by at least 50% reduction in baseline daily number of cigarettes
Smoking cessation service use | 3-month after baseline
  Any access to a smoking cessation service
Smoking cessation service use | 6-month after baseline
  Any access to a smoking cessation service
Use of nicotine replacement therapy | 3-month after baseline
  Any use of nicotine replacement therapy
Use of nicotine replacement therapy | 6-month after baseline
  Any use of nicotine replacement therapy
Change in nicotine dependence | 3-month after baseline
  Assessed by Heaviness of Smoking Index (range 0 to 6 with higher score indicating greater nicotine dependence)
Change in nicotine dependence | 6-month after baseline
  Assessed by Heaviness of Smoking Index (range 0 to 6 with higher score indicating greater nicotine dependence)
Number of quit attempt | 3-month after baseline
  Defined by abstinence for at least 24 hours
Number of quit attempt | 6-month after baseline
  Defined by abstinence for at least 24 hours
Intention to quit | 3-month after baseline
  Defined by readiness to quit in 30 days
Intention to quit | 6-month after baseline
  Defined by readiness to quit in 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Luk TT, Lam TH, Leung WC, Leung KY, Cheung KW, Kwa C, Siong KH, Tang KK, Lee KW, Hsieh CJ, Wu YS, Li WH, Wang MP. Brief Advice, Nicotine Replacement Therapy Sampling, and Active Referral for Expectant Fathers Who Smoke Cigarettes: A Randomized Clinical Trial. JAMA Intern Med. 2021 Aug 1;181(8):1081-1089. doi: 10.1001/jamainternmed.2021.2757. PMID 34125135
- [Derived] Luk TT, Hsieh CJ, Leung WC, Leung KY, Cheung KW, Kwa C, Siong KH, Tang KK, Lee KW, Li WH, Lam TH, Wang MP. Brief cessation advice, nicotine replacement therapy sampling and active referral (BANSAR) for smoking expectant fathers: Study protocol for a multicentre, pragmatic randomised controlled trial. Contemp Clin Trials. 2020 Jun;93:106006. doi: 10.1016/j.cct.2020.106006. Epub 2020 Apr 19. PMID 32320843